CLINICAL TRIAL: NCT05384886
Title: New Variants and Vaccines; Did it Cause a Change in the Mortality of COVID-19?
Brief Title: Impact of New Variants and Vaccines on the Course of COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Adnan Yamanoğlu, Assistant professor, Izmir Katip Celebi University
Other Study IDs: IRB-867
Record Dates: First submitted 2022-05-19; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; COVID-19 vaccines; SARS-CoV-2 strains; mortality; Case fatality rate
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1: COVID-19 patients in 2020: All patients over the age of 18 diagnosed with COVID-19 in 2020
  Interventions: Diagnostic Test: Polymerase chain reaction
- Group: COVID-19 patients in 2022: All patients over the age of 18 diagnosed with COVID-19 in 2022
  Interventions: Diagnostic Test: Polymerase chain reaction

INTERVENTIONS:
Diagnostic Test: Polymerase chain reaction — Covid-19 genetic material detection from mouth and nose swab

SUMMARY:
Novel coronavirus disease (COVID-19), caused by Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) virus, was first reported in December 2019 in Wuhan, China. The disease has spread to many countries in a few weeks and has become a global public health problem. By 2022, the virus has infected more than 500 million people worldwide and caused more than 6 million deaths.

Case fatality rates (CFR) are an important index that helps to understand the epidemiological characteristics of an epidemic. In the data coming in 2020, COVID-19 CFR values were generally reported in the range of 0.001-0.706. However, from 2019 to 2022, there were 2 major changes that could affect the CFR of the disease. The first of these is vaccine applications, and the second is the new variants of SARS-CoV-2, which appeared first. From 2019 to 2022, it is likely that there will be a change in the mortality of COVID-19 in relation to both the vaccines administered and the new variants emerging. However, the data on this subject are not clear yet and more studies are needed.

The aim of this study is to determine whether there is a change in the mortality of COVID-19 from 2019, when it first appeared, to 2022.

DETAILED DESCRIPTION:
Novel coronavirus disease (COVID-19), caused by Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) virus, was first reported in December 2019 in Wuhan, China. The disease spread to many countries in a few weeks, becoming a global public health problem, and the World Health Organization declared it a pandemic on March 11, 2020. COVID-19 has caused widespread deaths worldwide, especially by causing widespread involvement in the lungs and Acute Respiratory Distress Syndrome. By 2022, the virus has infected more than 500 million people worldwide and caused more than 6 million deaths.

Case fatality rates (CFR) are an important index that helps to understand the epidemiological characteristics of an epidemic. The CFR for COVID 19 is the number of deaths in COVID-19 cases divided by the total number of people infected with COVID-19. After the emergence of the disease in 2019, the CFR figures reported for COVID-19 in 2020 began to become clear. In the data coming in 2020, COVID-19 CFR values are generally reported in the range of 0.001-0.706. However, from 2019 to 2022, there were 2 major changes that could affect the CFR of the disease. The first of these is the vaccine applications developed against COVID-19. The first vaccine studies have matured by 2020 and started to be applied widely in the world in 2021. the second is the new variants of the first emerging SARS-CoV-2. In 2021, variants started to be defined and Alpha, Beta, Delta, and Omicron variants were reported as dominance variants from time to time. From 2019 to 2022, it is likely that there will be a change in the mortality of COVID-19 in relation to both the vaccines administered and the new variants emerging. Knowing the possible changes that may occur in COVID-19 mortality may cause changes in the COVID-19 measures applied all over the world. In this way, it may be possible to reduce unnecessary health costs and direct health resources to appropriate areas.

The aim of this study is to determine whether there is a change in the mortality of COVID-19 from 2019, when it first appeared, to 2022.

In this study, patient data were obtained retrospectively in a training and research hospital COVID-19 outpatient clinic. The obtained daily number of patients in 2020, CFR rates were compared with the number of daily patients and CFR rates in 2022. In this way, it was tested whether there was a significant difference between the year 2020, when the disease first became widespread, and 2022.

ELIGIBILITY:
Inclusion Criteria:

- All patients with a confirmed diagnosis of COVID-19 by PCR testing

Exclusion Criteria:

* Under 18 years old
* Clinical outcome cannot be followed
* Patients with severe trauma

Age Groups: Child, Adult, Older Adult
Study Population: All nontraumatic adult patients of both sexes with positive PCR tests and admitted with suspected symptoms of COVID-19 were included in the study.
Sampling Method: Probability Sample
Enrollment: 15967 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Number of COVID-19 patients diagnosed daily | 374 day
  Patients who applied to the COVID-19 outpatient clinic and service and whose diagnosis was confirmed by PCR test

SECONDARY OUTCOMES:
Case fatality rate | 374
  The ratio of the number of deaths in diagnosed cases to the total number of people infected.

CONTACTS AND LOCATIONS:
Locations (1):
- IKCU, Atatürk Eğitim ve Araştırma Hastanesi, Acil Tıp, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All data and statistical analyzes will be shared with academics and official institutions requesting the patient's names, provided that they remain confidential, after the permission of the institution.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting in January 2024